CLINICAL TRIAL: NCT03091868
Title: A Double-blind, Randomised, Placebo-controlled Study in Healthy Volunteers to Investigate the Tolerability and Pharmacokinetics of Rising Single-doses of BIA 6-512 and Their Effect on the Levodopa Pharmacokinetics When Administered in Combination With a Single-dose of Levodopa/Carbidopa 100/25 mg or With a Single-dose of Levodopa/Carbidopa 100/25 mg Plus a Single-dose of Entacapone 200 mg
Brief Title: Pharmacokinetics of Rising Single-doses of BIA 6-512 and Their Effect on the Levodopa Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-6512-102
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — entacapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (BIA 6-512 25 mg + Placebo) (Experimental): Single-doses were prepared as follows:
  BIA 6-512 25 mg dose = 1 capsule of 25 mg plus 1 capsule of placebo In all groups, placebo recipients received 2 capsules of placebo. BIA 6-512/Placebo capsules and Sinemet® 100/25 and Comtan® tablets were administered simultaneously, by oral route, in fasting conditions.
  Interventions: Drug: Placebo oral capsule; Drug: Sinemet® 100/25; Drug: Comtan®; Drug: BIA 6-512 25 mg
- Group 2 (BIA 6-512 50 mg + Placebo) (Experimental): Single-doses were prepared as follows:
  BIA 6-512 50 mg dose = 2 capsules of 25 mg In all groups, placebo recipients received 2 capsules of placebo. BIA 6-512/Placebo capsules and Sinemet® 100/25 and Comtan® tablets were administered simultaneously, by oral route, in fasting conditions.
  Interventions: Drug: Placebo oral capsule; Drug: Sinemet® 100/25; Drug: Comtan®; Drug: BIA 6-512 25 mg
- Group 3 (BIA 6-512 100 mg + Placebo) (Experimental): Single-doses were prepared as follows:
  BIA 6-512 100 mg dose = 1 capsule of 100 mg plus 1 capsule of placebo In all groups, placebo recipients received 2 capsules of placebo. BIA 6-512/Placebo capsules and Sinemet® 100/25 and Comtan® tablets were administered simultaneously, by oral route, in fasting conditions.
  Interventions: Drug: Placebo oral capsule; Drug: Sinemet® 100/25; Drug: Comtan®; Drug: BIA 6-512 100 mg
- Group 4 (BIA 6-512 200 mg + Placebo) (Experimental): Single-doses were prepared as follows:
  BIA 6-512 200 mg dose = 2 capsules of 100 mg In all groups, placebo recipients received 2 capsules of placebo. BIA 6-512/Placebo capsules and Sinemet® 100/25 and Comtan® tablets were administered simultaneously, by oral route, in fasting conditions.
  Interventions: Drug: Placebo oral capsule; Drug: Sinemet® 100/25; Drug: Comtan®; Drug: BIA 6-512 100 mg

INTERVENTIONS:
Drug: Placebo oral capsule — Matching placebo capsules. Oral administration.
Drug: Sinemet® 100/25 — Single-dose of immediate release levodopa/carbidopa 100/25 mg consisted of 1 tablet of Sinemet® 100/25. Route of administration: Oral.
Drug: Comtan® — Single-dose of entacapone 200 mg consisted of 1 tablet of Comtan®. Route of administration: Oral.
Drug: BIA 6-512 25 mg — BIA 6-512 capsules strengths 25 mg. Oral administration.
  Arms: Group 1 (BIA 6-512 25 mg + Placebo); Group 2 (BIA 6-512 50 mg + Placebo)
Drug: BIA 6-512 100 mg — BIA 6-512 capsules strengths 100 mg. Oral administration.
  Arms: Group 3 (BIA 6-512 100 mg + Placebo); Group 4 (BIA 6-512 200 mg + Placebo)

SUMMARY:
To investigate the effect of rising oral single-doses of BIA 6-512 (25 mg, 50 mg, 100 mg and 200 mg) on levodopa pharmacokinetics when administered in combination with a single-dose of immediate release levodopa/carbidopa 100/25 mg (Sinemet® 100/25) or with a single-dose of Sinemet® 100/25 plus a single-dose of entacapone (Comtan®) 200 mg and to assess the tolerability and safety of rising single oral doses of BIA 6-512 when administered in combination with a single-dose of Sinemet® 100/25 or with a single-dose of Sinemet® 100/25 plus a single-dose of Comtan® 200 mg.

DETAILED DESCRIPTION:
Single centre, double-blind, randomised, placebo-controlled study in four sequential groups of healthy subjects. Eligible subjects were admitted to the UFH on the day prior to receiving the first study medication. On the morning of the first dosing day (Day 1), subjects received BIA 6-512/Placebo concomitantly with Sinemet® 100/25; on the morning of the second dosing day (Day 2), subjects received BIA 6-512/Placebo concomitantly with Sinemet® 100/25 and Comtan® 200 mg. Products were administered in fasting conditions (at least 8 hours). Subjects remained confined in the UFH from admission (Day 0) until at least 24 h post last dose (Day 3); then, they were discharged and will return for the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Subjects who had clinical laboratory tests clinically acceptable at screening and admission.
* Subjects who had negative tests for HBsAg, anti-HCVAb and anti-HIV-1 and anti-HIV-2 Ab at screening.
* Subjects who had a negative screen for alcohol and drugs of abuse at screening and admission.
* Subjects who were non-smokers or who smoked less than 10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.
* (If female) She was sterile or, if of childbearing potential, she used one of the following methods of contraception: double barrier, intrauterine device or abstinence.
* (If female) She had a negative urine pregnancy test at screening and admission.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria, OR
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 21 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening or admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening or admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who had used prescription or over-the-counter medication within 2 weeks of admission.
* Subjects who had used any investigational drug or participated in any clinical trial within 3 months prior to screening.
* Subjects who had donated or received any blood or blood products within 3 months prior to screening.
* Subjects who were vegetarians, vegans or have medical dietary restrictions.
* Subjects who cannot communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not use an approved effective contraceptive method or she used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2004-11-03 (Actual); Primary Completion 2005-02-28 (Actual); Study Completion 2005-02-28 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) - Day 1 | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  Pharmacokinetic parameters for BIA 6-512, levodopa, 3-O-methyldopa (3-OMD) on Day 1 - Day of administration of BIA 6-512/Placebo concomitantly with 1 tablet of levodopa/carbidopa 100/25 mg (Sinemet® 100/25)
Time at which the Cmax occurred (tmax) - Day 1 | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  Pharmacokinetic parameters for BIA 6-512, levodopa, 3-O-methyldopa (3-OMD) on Day 1 - Day of administration of BIA 6-512/Placebo concomitantly with 1 tablet of levodopa/carbidopa 100/25 mg (Sinemet® 100/25)
Area under the plasma concentration versus time curve (AUC) from time zero to the last sampling time at which concentrations were at or above the limit of quantification (AUC0-t) - Day 1 | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  Pharmacokinetic parameters for BIA 6-512, levodopa, 3-O-methyldopa (3-OMD) on Day 1 - Day of administration of BIA 6-512/Placebo concomitantly with 1 tablet of levodopa/carbidopa 100/25 mg (Sinemet® 100/25)
AUC from time zero to the infinity (AUC0-∞) - Day 1 | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  Pharmacokinetic parameters for BIA 6-512, levodopa, 3-O-methyldopa (3-OMD) on Day 1 - Day of administration of BIA 6-512/Placebo concomitantly with 1 tablet of levodopa/carbidopa 100/25 mg (Sinemet® 100/25)
Elimination rate constant (λz) - Day 1 | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  Pharmacokinetic parameters for BIA 6-512, levodopa, 3-O-methyldopa (3-OMD) on Day 1 - Day of administration of BIA 6-512/Placebo concomitantly with 1 tablet of levodopa/carbidopa 100/25 mg (Sinemet® 100/25)
Apparent elimination half-life (t1/2) - Day 1 | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  Pharmacokinetic parameters for BIA 6-512, levodopa, 3-O-methyldopa (3-OMD) on Day 1 - Day of administration of BIA 6-512/Placebo concomitantly with 1 tablet of levodopa/carbidopa 100/25 mg (Sinemet® 100/25)
Maximum observed plasma drug concentration (Cmax) - Day 2 | ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  Pharmacokinetic parameters for BIA 6-512, levodopa, 3-O-methyldopa (3-OMD) and entacapone on day 2 - Day of administration of BIA 6-512/Placebo concomitantly with 1 tablet of levodopa/carbidopa 100/25 mg (Sinemet® 100/25) plus 1 tablet of entacapone 200 mg (Comtan®). Administration occurred 24 h after the time of administration in Day 1.
Time at which the Cmax occurred (tmax) - Day 2 | ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  Pharmacokinetic parameters for BIA 6-512, levodopa, 3-O-methyldopa (3-OMD) and entacapone on day 2 - Day of administration of BIA 6-512/Placebo concomitantly with 1 tablet of levodopa/carbidopa 100/25 mg (Sinemet® 100/25) plus 1 tablet of entacapone 200 mg (Comtan®). Administration occurred 24 h after the time of administration in Day 1.
Area under the plasma concentration versus time curve (AUC) from time zero to the last sampling time at which concentrations were at or above the limit of quantification (AUC0-t) - Day 2 | ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  Pharmacokinetic parameters for BIA 6-512, levodopa, 3-O-methyldopa (3-OMD) and entacapone on day 2 - Day of administration of BIA 6-512/Placebo concomitantly with 1 tablet of levodopa/carbidopa 100/25 mg (Sinemet® 100/25) plus 1 tablet of entacapone 200 mg (Comtan®). Administration occurred 24 h after the time of administration in Day 1.
AUC from time zero to the infinity (AUC0-∞) - Day 2 | ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  Pharmacokinetic parameters for BIA 6-512, levodopa, 3-O-methyldopa (3-OMD) and entacapone on day 2 - Day of administration of BIA 6-512/Placebo concomitantly with 1 tablet of levodopa/carbidopa 100/25 mg (Sinemet® 100/25) plus 1 tablet of entacapone 200 mg (Comtan®). Administration occurred 24 h after the time of administration in Day 1.
Elimination rate constant (λz) - Day 2 | ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  Pharmacokinetic parameters for BIA 6-512, levodopa, 3-O-methyldopa (3-OMD) and entacapone on day 2 - Day of administration of BIA 6-512/Placebo concomitantly with 1 tablet of levodopa/carbidopa 100/25 mg (Sinemet® 100/25) plus 1 tablet of entacapone 200 mg (Comtan®). Administration occurred 24 h after the time of administration in Day 1.
Apparent elimination half-life (t1/2) - Day 2 | ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  Pharmacokinetic parameters for BIA 6-512, levodopa, 3-O-methyldopa (3-OMD) and entacapone on day 2 - Day of administration of BIA 6-512/Placebo concomitantly with 1 tablet of levodopa/carbidopa 100/25 mg (Sinemet® 100/25) plus 1 tablet of entacapone 200 mg (Comtan®). Administration occurred 24 h after the time of administration in Day 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Pharmacology Unit (UFH), S. Mamede Do Coronado, Portugal

IPD SHARING:
Plan to Share IPD: Undecided